CLINICAL TRIAL: NCT03663556
Title: Feeding the Preterm Gut Microbiota - Impact of Infant-feeding on Preterm Gut Microbiota Development
Acronym: FEEDMI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universidade do Porto (Other)
Collaborators: Center for Health Technology and Services Research (Other); Maternidade Dr. Alfredo da Costa (Unknown); Universidade Nova de Lisboa (Other)
Responsible Party: Sponsor
Other Study IDs: FEEDMI
Record Dates: First submitted 2018-07-19; First posted 2018-09-10 (Actual); Last update posted 2018-10-02 (Actual); Status verified 2018-08

CONDITIONS: Very Preterm Infants
Keywords: intestinal microbiota; preterm infants; breast milk; donor human milk; formula

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Meconium and stool samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Very Preterm Infants: Newborn infants with less than 32 weeks admitted in the NICU.
  Interventions: Other: Infant-feeding

INTERVENTIONS:
Other: Infant-feeding — Preterm infants hospitalized in the NICU can be feed by three different types of infant feeding, such as breast milk, donor human milk and/or formulas.

SUMMARY:
Preterm infants are especially vulnerable to gut microbiota disruption and dysbiosis since their early gut microbiota is less abundant and diverse. Several factors may influence infants' microbiota such as mother's diet, mode of delivery, antibiotic exposure and type of feeding. The main goal of this observational study is to evaluate the impact of different types of feeding (breast milk, donor human milk and preterm formulas) on the intestinal microbiota of preterm infants hospitalized in the neonatal intensive care unit (NICU) of Maternidade Alfredo da Costa (MAC). Furthermore, the influence of mode of delivery and the mother's diet, among others factors, on vertical microbiota transmission will be evaluated. After delivery, mothers will be asked to collect their own fecal samples and will be invited to complete a semi-quantitative food frequency questionnaire. Stool samples will be collected from premature infants every 7 days. DNA will be extracted from fecal samples and different bacterial genus and species will be analyzed.

DETAILED DESCRIPTION:
Meconium and the additional 3 fecal samples will be collected from preterm infants by the nursing team of MAC Neonatology Unit. Fecal samples will be collected every 7 days, during 21 days, from diapers into sterile tubes. Mothers will be asked to collect their own fecal samples with an appropriate stool collection kit (EasySampler®) and will be invited to complete a semi-quantitative food frequency questionnaire, previously validated for the Portuguese population.

Infant-feeding profile (breast milk, donor human milk or formula) of preterm infants will be recorded every day to select the most representative (>50 %) type of infant-feeding received during the 7 days prior to each fecal sample collection.

Additionally, detailed clinical data will be collected during the preterm infant enrollment in the study. Personal clinical data includes sociodemographic information and clinical intrapartum and postpartum outcomes, such as newborn's weight, days of antibiotic exposure, number of total days of hospitalization and others outcomes related to the preterm clinical evolution.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible for enrolment, preterm infants must have been admitted to the NICU in less than 24 hours of life, have been born with less than 32 weeks with absence of malformations or metabolic diseases.

Exclusion Criteria:

* non applicable

Max Age: 2 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Very preterm infants born with less than 32 weeks recruited at the NICU of Maternidade Dr. Alfredo da Costa, Centro Hospitalar de Lisboa Central, Lisbon, Portugal
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2017-05-25 (Actual); Primary Completion 2018-12-30 (Estimated); Study Completion 2018-12-30 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline intestinal microbiota composition of preterm infants at 7, 14 and 21 days. | The first fecal sample (meconium) of preterm infants will be collected. Afterwards, fecal samples will be collected every 7 days, during 21 days.
  The intestinal microbiota profile of preterm infants will be evaluated over time.
Changes from baseline intestinal microbiota composition of preterm infants in relation to infant-feeding profile (breast milk, donor human milk or formula) at 7,14 and 21 days. | Infant-feeding type of preterm infants before the first, second, third and fourth collection will be recorded during these 21 days.
  Infant-feeding profile (breast milk, donor human milk or formula) will be recorded every day to select the most representative type of infant-feeding (> 50 %) received during the 7 days prior to each fecal sample collection.

SECONDARY OUTCOMES:
Maternal intestinal microbiota composition, analyzed by RT-PCR. | Maternal fecal samples will be collected after delivery up to 1 week.
  Mother's will be asked to collect their own fecal samples for gut microbiota analysis by RT-PCR. An appropriate stool collection kit will be provided (EasySampler Stool Collection kit).
Changes in maternal gut microbiota in relation to clinical variables described below | Clinical variables will be collected daily, until study completion an average of 2 years.
  Changes in intestinal microbiota profile of preterm infants' mothers will be evaluated in relation to mode of delivery, mother's gestational age, dietary pattern during pregnancy, weight gain in gestation and antibiotic exposure.

CONTACTS AND LOCATIONS:
Locations (2):
- Portugal (2):
  - Maternidade Dr. Alfredo da Costa, Centro Hospitalar de Lisboa Central, Lisbon
  - NOVA Medical School, Universidade Nova de Lisboa, Lisbon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Morais J, Marques C, Teixeira D, Durao C, Faria A, Brito S, Cardoso M, Macedo I, Pereira E, Tome T, Calhau C. Extremely preterm neonates have more Lactobacillus in meconium than very preterm neonates - the in utero microbial colonization hypothesis. Gut Microbes. 2020 Nov 9;12(1):1785804. doi: 10.1080/19490976.2020.1785804. Epub 2020 Jul 13. PMID 32658601